CLINICAL TRIAL: NCT04361591
Title: COVID-19 in Liver Transplant Recipients in Spain: a Nationwide Prospective Study
Brief Title: COVID-19 in Liver Transplant Recipients
Acronym: COVID19-SETH
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Sociedad Española de Trasplante Hepático (Network)
Responsible Party: Principal Investigator, Jordi Colmenero, Liver Transplant Hepatologist, SETH Scientific Committee Chair, Hospital Clinic of Barcelona
Other Study IDs: HCB/2020/0384
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Liver Transplant; Complications; COVID19; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Liver Transplant recipients
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — Observational Study

SUMMARY:
Prospective observational study aimed at analyzing the incidence, clinical characteristics and outcomes of COVID-19 in LT in Spain.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is a novel viral disease caused by the SARS-Cov-2 infection with a particular predominance of upper and lower respiratory tract symptoms. First diagnosed in China in late 2019, the virus has progressed to a state of pandemia, involving Spain with a important outbreak.

While the outcomes of viral infections in solid organ transplant (SOT) recipients tend to be worse than those from the general population due to chronic immunosuppression, there is little information on the incidence and outcomes of COVID-19 in liver transplant (LT) recipients. LT recipients are usually under less immunosuppression than other SOT and the clinical expression and outcomes of COVID-19 may be different to the reported outcomes in other SOT.

The Spanish Society of Liver Transplantation, which includes 25 LT programs, has promoted a nationwide registry for LT with COVID-19 to help ascertain the incidence and outcomes and help evidence-based management .

ELIGIBILITY:
Inclusion Criteria:

* Liver Transplant recipient
* Confirmed (PCR positive) SARS-Cov-2 infection
* Informed Consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Liver Transplantation
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID19 in LT recipients | 12 months
Clinical characteristics of COVID19 in LT recipients | 12 months
Survival and Mechanical ventilation / respiratory support | 3 months
Observed treatments and immunosuppression management | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Colmenero, Principal Investigator — Sociedad Española de Trasplante Hepático
Locations (1):
- SETH-affiliated Liver Transplant Programs in Spain, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SETH webpage — https://www.sethepatico.org/